CLINICAL TRIAL: NCT06277362
Title: "Arterial-Venous Reversal Flow in "No-option" Chronic Limb-threating Ischemia (CLTI) Patients"
Brief Title: Peripheral Extreme Revascularization in "No-option" Patiens With Chronic Limb Threatening Ischemia
Acronym: PiPER
Status: Recruiting | Type: Observational
Sponsor: EndoCore Lab s.r.l. (Other)
Responsible Party: Sponsor
Other Study IDs: CLTI012023
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease; Critical Limb-Threatening Ischemia; Diabetic Foot
Keywords: PAD; DVA; CLTI
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to evaluate early safety and effectiveness of the percutaneous deep foot venous arterialization performed in clinical practice, in an unselected population of patients with "no-option" CLTI.

DETAILED DESCRIPTION:
Critical lower Limb Threatening Ischemia is the most advanced stage of lower limb arterial disease and is associated with a high risk of mortality and major amputation.Literature data indicate that about 5-10% of patients with peripheral arterial disease have a risk of developing CLTI, therefore the most advanced stage of arterial disease of the lower limbs, within 5 years and have a mortality of 20% at 6 months after diagnosis of CLTI.Despite the continuous improvement of the techniques and materials used in the revascularization of these patients, the data of the Literature show that in about 10-15% of these patients revascularization is impossible or ineffective. This condition is defined as: "no-option" CLTI.Therefore, for patients with "no-option" CLTI an alternative treatment for limb rescue may be considered the use of arterialization of the venous plexus of the foot; that is, to use to bring the arterial flow to the foot a healthy conduit, such as the vein, instead of the diseased artery and no longer usable.

The present study is designed as a multicentre, prospective, single-arm, observational study.

All eligible subjects for undergoing PiPER procedure at sites participating in the study will be considered for enrolment and will be asked to give consent prior to participating.

Subjects will be considered enrolled in the study at the time written informed consent is given to the use of their personal data. Once patients are enrolled, their demographics, medical history, disease-relevant conditions, treatment details and outcomes will be collected for up to 24 months from the procedure.

The study will collect information about the medical care patients receive during their planned procedure. No additional testing or procedures will be done.

The revascularization procedure will be performed as per the current clinical practice.

After discharge all patients will attend clinic visits at 30 days (±7 days), 6 months (±14 days),12 months (±30 days), 24 months (±30 days).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient has signed an approved informed consent form
* All patients, with non-revascularizable critical lower limb ischemia defined on the basis of 2 previous unsuccessful Percutaneous Transluminal Angioplasty (PTA) attempts or on severe Medial Artery Calcification (MAC)/Small Artery Disease (SAD) stage.
* Patient with Critical Limb Ischaemia, Rutherford category, 5 (minor tissue loss) or 6 (major tissue loss) with active trophic lesions
* Ejection Fraction > 30%

Exclusion Criteria:

* Subject no able to perform the follow up or other factors making clinical follow-up difficult
* Patients with critical ischaemia of the lower limbs revascularizable by bypass or angioplasty, critical ischaemia characterised by rest pain (Rutherford class ≤ 4)
* Ejection Fraction < 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting the most advanced stage of lower limb arterial disease, defined as patients with CLTI and no indication for revascularization.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety Composite | 30 days, 6 months
  Composite of amputation free survival, defined as the rate of limb salvage (freedom from major amputation) and survival (freedom from all causes of death) of the percutaneous deep foot venous arterialization procedure.

SECONDARY OUTCOMES:
Procedural Success | Day 1
  Procedural success (defined as completion of the procedure by percutaneous route with achievement of arterial flow in the venous plexus of the foot at the end, as angiographically assessed);
Primary Patency | 30 days, 3 months, 6 months, 12 months and 24 months
  Primary patency defined as no occlusion of the arterialized vein tract
Secondary Patency | 30 days, 3 months, 6 months, 12 months and 24 months
  Secondary patency defined as no secondary occlusion of the arterialised vein tract
A-V fistula flow rate | 30 days, 3 months, 6 months, 12 months and 24 months
  A-V fistula flow rate
Minor amputation rates | 30 days, 3 months, 6 months, 12 months and 24 months
  Minor amputation rates defined as a below the ankle amputation
Major amputation rates | 30 days, 3 months, 6 months, 12 months and 24 months
  Major amputation rates defined as an above the ankle amputation
Re-Treatment rate | 30 days, 3 months, 6 months, 12 months and 24 months
  Re-Treatment rate defined as need for reintervention
Wound Size | Baseline, 30 days, 3 months, 6 months, 12 months and 24 months
  Wound Size defined as wound size reduction index
TpcO2 | Baseline, 30 days, 3 months, 6 months, 12 months and 24 months
  TpcO2 defined as TpcO2 value changes
WIFi class | Baseline, 30 days, 3 months, 6 months, 12 months and 24 months
  WIFi class and stage changes
Freedom from all cause death | 30 days, 3 months, 6 months, 12 months and 24 months
  Freedom from all cause death
Freedom from procedure-related death | 30 days, 3 months
  Freedom from procedure-related death
Rutherford class | Baseline, 30 days, 3 months, 6 months, 12 months and 24 months
  Rutherford class and stage changes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Morselli, PharmD, Study Director — EndocoCore Lab s.r.l.; Bruno Migliara, MD, Principal Investigator — Casa di Cura Pederzoli; Marco Manzi, MD, Study Chair — Casa di Cura Abano Terme
Locations (7):
- Italy (7):
  - Ospedale Pederzoli, Peschiera del Garda, Veneto
  - Ospedale San Martino, Belluno
  - Ospedale Bufalini, Cesena
  - Ospedale di Conegliano - USLL2, Conegliano
  - Ospedale Cardarelli, Napoli
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale Santa Chiara, Trento